CLINICAL TRIAL: NCT04935515
Title: C Reactive Protein Based Early Intervention for Home Quarantined COVID -19 Patients to Avoid Complications and Hospitalization.
Brief Title: C Reactive Protein in Home Quarantined Coronavirus Disease 2019 (COVID -19) Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manimarane Arjunan, MD,DM (Cardiology) (Other)
Collaborators: UR Anoop Research Group (Other)
Responsible Party: Sponsor-Investigator, Manimarane Arjunan, MD,DM (Cardiology), Principal Investigator, UR Anoop Research Group
Organization: UR Anoop Research Group (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1/MA/URA/21
Record Dates: First submitted 2021-06-20; First posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: COVID -19
Keywords: COVID -19;; Home quarantine;; C-Reactive Protein (CRP);; D-Dimer,; Early Intervention prior to onset of hypoxia
MeSH Terms: conditions — COVID-19 | interventions — Anti-Bacterial Agents; Histamine Antagonists; Anti-Inflammatory Agents; Geritol; Steroids; Anticoagulants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mild (Experimental): Patients with mild symptoms and normal CRP.
  Interventions: Drug: Oral Antibiotic, Antihistamine, Anti-inflammatory, Multivitamins
- Moderate (Experimental): Patients with mild symptoms and less than 10 fold increase in CRP.
  Interventions: Drug: Oral Antibiotic, Antihistamine, Anti-inflammatory, Multivitamins; Drug: Oral low dose steroid; Drug: Oral anti-coagulant
- Severe (Experimental): Patients with high grade fever persisting even on the third or fourth day after onset of symptoms or 10 fold or more increase in CRP.
  Interventions: Drug: Intravenous Antibiotics with Low dose steroid.; Drug: Oral anti-coagulant

INTERVENTIONS:
Drug: Oral Antibiotic, Antihistamine, Anti-inflammatory, Multivitamins — Oral Azithromycin , Cetirizine, Paracetamol, Zinc, Vitamin C, Vitamin D
  Arms: Mild; Moderate
Drug: Oral low dose steroid — Low dose oral methyl prednisolone was added.
  Arms: Moderate
Drug: Intravenous Antibiotics with Low dose steroid. — Intravenous ceftriaxone with either oral methyl prednisolone or intravenous dexamethasone was given
  Arms: Severe
Drug: Oral anti-coagulant — Rivaroxaban was given for minimum 4 weeks depending on D dimer levels
  Arms: Moderate; Severe

SUMMARY:
During the peak of the second COVID -19 wave, the hospitals were over-crowded. Many COVID -19 positive patients had to stay at home and reach out to their family physicians for guidance. Medical follow-up for these patients was a daunting challenge. As in - patient hospital facilities were not readily accessible due to over crowding, early objective tests to identify home quarantined patients prone to deterioration and timely medical intervention to avoid hospitalization were required.

Based on early assessment of inflammatory markers like CRP and clinical signs like persistent high-grade fever, need-based early medical intervention was initiated in home quarantined COVID -19 patients prior to the onset of hypoxia, in order to avoid complications and hospitalization

DETAILED DESCRIPTION:
25 home quarantined COVID -19 patients who contacted online for medical guidance underwent clinical and biochemical evaluation. Radiological evaluation was done only if indicated.

Based on early objective biochemical tests like elevated CRP and clinical signs like persistent high-grade fever on the third or fourth day after onset of symptoms, early medical treatment was initiated prior to onset of hypoxia.

All the 25 patients recovered without any complications and did not require hospitalization.

ELIGIBILITY:
Inclusion Criteria:

1. COVID -19 positive patients under home quarantine
2. Patients consulting online on the 3rd or 4th day after the onset of symptoms.
3. Patients with oxygen saturation 94% and above.

Exclusion Criteria:

1. Patients consulting online on or after 5th day of onset of symptoms.
2. Patients with oxygen saturation less than 94% during the initial presentation.
3. Systemic disease known to increase CRP levels.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-05-09 (Actual); Study Completion 2021-06-06 (Actual)

PRIMARY OUTCOMES:
Number of home quarantined COVID -19 positive patients requiring admission in a hospital for hypoxia. | Two weeks from the onset of symptoms.
  Oxygen saturation in COVID-19 positive patients was monitored using pulse oximetry at home. Those patients who developed hypoxia (less than 94%) were referred for hospitalization.

SECONDARY OUTCOMES:
Number of home quarantined COVID -19 patients developing thromboembolic complications | Four weeks from the time of initial presentation
  Thromboembolic complications in COVID-19 positive patients under home quarantine were assessed using an online questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: MANIMARANE ARJUNAN, MD,DM-CARDIO, Principal Investigator — UR Anoop Research Group
Locations (1):
- ONLINE, Puducherry, India

IPD SHARING:
Plan to Share IPD: No